CLINICAL TRIAL: NCT03674125
Title: A Multi-center, Open-label, Dose-ranging, Phase 1 Study to Evaluate the Safety, Tolerability, and Immunogenicity of GLS-6150, Administered ID and Followed by Cellectra® 2000 Healthy Adults and in Persons Previously Treated for Hepatitis C Virus Infection.
Brief Title: Evaluation of Safety, Tolerability, and Immunogenicity Study of GLS-6150 in Healthy Volunteers and in Persons Previously Treated for Hepatitis C Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GeneOne Life Science, Inc. (Industry)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCV-003
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: HCV Infection
Keywords: Hepatitis C Virus; HCV; Vaccine; DNA
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): GLS-6150 at 2.0 mg DNA/dose (3 dose prime plus boost)
  Interventions: Biological: GLS-6150
- Group 2 (Experimental): GLS-6150 at 1.0 mg DNA/dose (3 dose prime plus boost)
  Interventions: Biological: GLS-6150
- Group 3 (Experimental): GLS-6150 at 2.0 mg DNA/dose(3 dose prime plus boost)
  Interventions: Biological: GLS-6150
- Group 4 (Experimental): GLS-6150 at 2.0 mg DNA/dose(2 dose prime plus boost)
  Interventions: Biological: GLS-6150

INTERVENTIONS:
Biological: GLS-6150 — Group 1: GLS-6150 2.0 mg at 0, 4, 12, and 24 weeks (N=8, healthy volunteers); Group 2: GLS-6150 1.0 mg at 0, 4, 12, and 24 weeks (N=8, previously treated for HCV infection); Group 3: GLS-6150 2.0 mg at 0, 4, 12, and 24 weeks (N=8, previously treated for HCV infection); Group 4: GLS-6150 2.0 mg at 0, 8, and 24 weeks (N=8, previously treated for HCV infection)

SUMMARY:
Hepatitis C virus (HCV) is an enveloped, single strand, positive sense RNA flavivirus. Infection by HCV is typically chronic, although an estimated ~10-20% may spontaneously clear the virus. HCV affects between 1.3 - 2 billion individuals, or 2-3% of the global population. HCV has a seroprevalence of approximately 1% in developed countries such as the US and Korea. Chronic HCV infection leads to hepatic fibrosis and cirrhosis. This Phase I study will evaluate the safety, tolerability and immunogenicity of GLS-6150 administered intradermally (ID) followed by electroporation at 1.0 mg and 2.0 mg/dose assessing 3 and 4-dose regimens.

DETAILED DESCRIPTION:
HCV-003 will assess the safety and immunogenicity of GLS-6150 in those previously treated for HCV infection and who have achieved a sustained virologic response (SVR). This study will provide information as to whether GLS-6150 may be useful to prevent re-infection for those successfully cleared of HCV infection. GLS-6150 is a DNA plasmid vaccine that expresses the NS3/4A gene of HCV, NS4B gene of HCV, the NS5A gene of HCV and IL-28B. GLS-6150 will be administered at one of two dose levels (1 mg or 2 mg) and given as a 2 or 3 vaccination priming regimen with a boost vaccination given at 6 months. Immune T cell and serologic responses will be determined after each dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-65 years;
2. HCV seronegative (Group 1 only), HCV seropositive (Groups 2, 3, 4 only)
3. Prior treatment for genotype 1a or 1b Hepatitis C infection with treatment ending (12 weeks after end of DAA treatment, 24 weeks after end of combination treatment with Ribavirin/Interferon) prior to study enrollment and with documented achievement of HCV viral clearance (multiple episodes of treatment for Hepatitis C are allowed, Groups 2, 3, 4 only)
4. Hepatitis C virus PCR negative at screen
5. Able to provide consent to participate and having signed an Informed Consent Form (ICF);
6. Able and willing to comply with all study procedures;
7. Women of child-bearing potential agree to use medically effective contraception (oral contraception, barrier methods, spermicide, etc.) or have a partner who is sterile during this trial, or have a partner who is medically unable to induce pregnancy.
8. Normal screening ECG or screening ECG with no clinically significant findings;
9. Screening laboratory must be within normal limits or have only Grade 0-1 findings;
10. No history of clinically significant immunosuppressive or autoimmune disease.
11. Not currently or within the previous 4 weeks taking immunosuppressive agents (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or prednisone at a dose less than 10 mg/day, or a steroid equivalent).

Exclusion Criteria:

1. Administration of an investigational compound either currently or within 3 months of first dose;
2. Administration of any vaccine (excluding influenza vaccination) within 4 weeks of first dose;
3. Administration of any monoclonal or polyclonal antibody product within 4 weeks of the first dose
4. Administration of any blood product within 3 months of first dose;
5. Pregnancy or breast feeding or plans to become pregnant during the course of the study;
6. History of positive serologic test for HIV, hepatitis B surface antigen (HBsAg); or any potentially communicable infectious disease as determined by the Principal Investigator or Medical Monitor;
7. Positive Hepatitis C serology performed at baseline (Group 1 only)
8. Positive screening PCR test for hepatitis C virus;
9. History of HCV infection with other than genotype 1a or 1b (Group 2, 3 and 4 only)
10. Baseline evidence of kidney disease as measured by creatinine greater than 1.5 mg/dL
11. Baseline screening lab(s) with Grade 2 or higher abnormality;
12. Chronic liver disease, cirrhosis, hemochromatosis, Wilson's disease, alcoholic liver disease, autoimmune hepatitis, or α-1 antitrypsin deficiency(In case of cirrhosis, the person who has been judged F4 grade in Fibroscan);
13. Immunosuppressive illness including hematologic malignancy, history of solid organ or bone marrow transplantation;
14. Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, low-dose methotrexate, or prednisone at a dose equal to or greater than 10 mg/day, or steroid equivalent);
15. Current or anticipated treatment with TNF-α inhibitors such as infliximab, adalimumab, etanercept;
16. Prior major surgery or any radiation therapy within 4 weeks of the first vaccination;
17. Any pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome; history of PSVT syndrome, history of prolonged QT syndrome;
18. Presence of a cardiac pacemaker or automatic implantable cardioverter defibrillator (AICD)
19. Metal implants within 20 cm of the planned site(s) of injection;
20. Presence of keloid scar formation or hypertrophic scar as a clinically significant medical condition at the planned site(s) of injection.
21. Prisoner or subjects who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness;
22. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints; or
23. Not willing to allow storage and future use of samples for Hepatitis C virus related research
24. Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Day0 through up to 28 weeks
Administration (injection) site reactions | Day0 through up to 28 weeks
Changes in safety laboratory parameters described by frequency and severity grade | Day0 through up to 28 weeks

SECONDARY OUTCOMES:
Antigen specific cellular immune responses to Hepatitis C virus as determined by Interferon-gamma (IFN-γ) ELISpot and/or FACS assay | Day0 through up to 28 weeks
Binding antibody titers to the HCV non-structural proteins (NS3, NS4, NS5) measured by ELISA | Day0 through up to 28 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Pusan National University Hospital, Busan
  - Yonsei University Health System, Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided